CLINICAL TRIAL: NCT05080933
Title: Extracorporeal Membrane Oxygenation for COVID-19 and Influenza H1N1 Associated Acute Respiratory Distress Syndrome: a Multi-centre Retrospective Cohort Study
Brief Title: ECMO for COVID-19 vs Influenza A H1N1 Associated ARDS
Acronym: InfluCOV_ECMO
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Vito Fanelli MD, PhD, MD, PhD, University of Turin, Italy
Other Study IDs: v1_12_2020
Record Dates: First submitted 2021-10-15; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: ARDS; COVID-19; H1N1 Influenza
MeSH Terms: conditions — COVID-19; Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19
- H1N1

SUMMARY:
Objective: Veno-venous ECMO has been used as a rescue therapy for patients with severe ARDS associated to influenza A H1N1 and COVID19 viral pneumonia. Little is known about outcome of these patients who required extracorporeal support.

Research question: To compare outcome of patients who required VV ECMO for Covid19 and H1N1 associated ARDS

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 or influenza A H1N1 (suspected or confirmed) diagnosis
* Severe ARDS (according to Berlin Definition)
* VV ECMO
* Invasive mechanical ventilation through endotracheal tube or tracheostomy

Exclusion Criteria:

• Age<18 years

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who required VV ECMO for COVID-19 and influenza A H1N1 associated ARDS
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2009-08-22 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
All cause mortality on day 60 after ECMO initiation | 60 days

SECONDARY OUTCOMES:
Hospital length of stay | 90 days
ICU length of stay | 90 days
Hospital mortality on day 90 after ECMO initiation | 90 days
ECMO duration | 90 days
ECMO associated hemorrhagic complications | 60 days
ECMO associated mechanical complications | 60 days
Invasive mechanical ventilation duration | 90 days
ECMO related haemorrhagic complications | 90 days
ECMO related mechanical complications | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fanelli V, Giani M, Grasselli G, Mojoli F, Martucci G, Grazioli L, Alessandri F, Mongodi S, Sales G, Montrucchio G, Pizzi C, Richiardi L, Lorini L, Arcadipane A, Pesenti A, Foti G, Patroniti N, Brazzi L, Ranieri V. Extracorporeal membrane oxygenation for COVID-19 and influenza H1N1 associated acute respiratory distress syndrome: a multicenter retrospective cohort study. Crit Care. 2022 Feb 5;26(1):34. doi: 10.1186/s13054-022-03906-4. PMID 35123562